CLINICAL TRIAL: NCT03042741
Title: Phase II Trial of Daily Dose of Oral Vaccine Against Atherosclerosis
Brief Title: Vaccine Against Atherosclerosis in Patients With Overweight Problems or Obesity
Acronym: V6
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Immunitor LLC (Industry)
Collaborators: Federal State Budget Institution Research Center for Obstetrics, Gynecology and Perinatology Ministry of Healthcare (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: V6
Record Dates: First submitted 2017-02-01; First posted 2017-02-03 (Estimated); Last update posted 2019-04-16 (Actual); Status verified 2018-08

CONDITIONS: Atherosclerosis
MeSH Terms: conditions — Atherosclerosis

STUDY DESIGN:
Intervention Model Description: Group on experimental drug compared against group receiving placebo in randomized, blinded phase III study to evaluate effect on lipid profile, i.e., LDL, HDL, triglycerides and total cholesterol
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-blind study in two groups of patients assigned randomly into experimental and placebo arms
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- V6 recipients (Experimental): Arm will comprise 150 individuals with overweight problem or obesity randomly assigned to receive V6 - oral atherosclerosis vaccine administered once per day for one month
  Interventions: Biological: atherosclerosis vaccine
- Placebo recipients (Placebo Comparator): Arm will comprise 150 individuals with overweight problem or obesity randomly assigned to receive placebo pills given once per day as a single pill for one month
  Interventions: Biological: Placebo pills

INTERVENTIONS:
Biological: atherosclerosis vaccine — Atherosclerosis vaccine, V6, formulated as an oral pill made from from pooled antigens derived from adipose tissue
  Arms: V6 recipients
Biological: Placebo pills — Half of the patients will be randomly assigned to receive placebo pill
  Arms: Placebo recipients

SUMMARY:
Atherosclerosis vaccine, V6, has been through two small-scale Phase II open label clinical trials. It has shown significant improvement in lipid profile in patients with overweight or obesity

DETAILED DESCRIPTION:
The proposed study will evaluate daily dose of one V6 pill administered for one month in placebo-controlled, randomized, double-blind phase 3 trial in men and women with baseline waist diameter over 90 and 80 cm respectively. The effect of V6 will be assessed by changes in lipid profile, i.e., LDL, HDL, TG and TC; anthropomorphic indices, i.e., circumference of waist, mid-arm, and hips; arterial blood pressure and fasting glucose levels at baseline versus post-treatment timepoint.

ELIGIBILITY:
Inclusion Criteria:

* Baseline waist diameter over 90 and 80 cm for men and women, respectively

Exclusion Criteria:

* Pregnant and lactating women
* Individuals with clinical symptoms or diseases who in opinion of study investigators are not eligible to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2017-02-01 (Actual); Primary Completion 2019-12-18 (Estimated); Study Completion 2019-12-18 (Estimated)

PRIMARY OUTCOMES:
Immunotherapy of atherosclerosis | 1 month
  Effect on lipid profile as measured by changes in LDL, HDL, triglycerides and total cholesterol

SECONDARY OUTCOMES:
Effect on anthropomorphic indices of obesity | 1 month
  Effect on diameter of waist, mid-arm and hip after one month of treatment versus baseline measurements
Effect on hypertension | 1 month
  The systolic and diastolic blood pressures measured one month apart
Effect on glucose levels | 1 month
  Changes in fasting glucose levels from baseline to post-treatment time-point

CONTACTS AND LOCATIONS:
Overall Officials: Allen Bain, PhD, Study Chair — Immunitor Inc.
Locations (1):
- Immunitor LLC, Ulaanbaatar, CA, Mongolia

IPD SHARING:
Plan to Share IPD: Undecided
Data will be shared without identification of participants

REFERENCES:
- [Background] Bourinbaiar AS, Jirathitikal V. Effect of oral immunization with pooled antigens derived from adipose tissue on atherosclerosis and obesity indices. Vaccine. 2010 Mar 24;28(15):2763-8. doi: 10.1016/j.vaccine.2010.01.032. Epub 2010 Jan 29. PMID 20117273
- [Background] Bourinbaiar AS, Jirathitikal V. Safety and efficacy trial of adipose-tissue derived oral preparation V-6 Immunitor (V-6): results of open-label, two-month, follow-up study. Lipids Health Dis. 2010 Feb 2;9:14. doi: 10.1186/1476-511X-9-14. PMID 20122177